CLINICAL TRIAL: NCT01962987
Title: A Randomized, Double-Blind, Multiple-Site, Placebo-Controlled, Parallel Design Study Comparing Diclofenac Sodium Gel 3% (Actavis) to Solaraze ® (Diclofenac Sodium) Gel 3% (Fougera Pharms) in the Treatment of Actinic Keratosis
Brief Title: A Study Comparing Diclofenac Sodium Gel 3% to Solaraze® (Diclofenac Sodium) Gel 3% in the Treatment of Actinic Keratosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 71204901
Record Dates: First submitted 2013-10-10; First posted 2013-10-16 (Estimated); Results first posted 2020-07-20 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — Diclofenac

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Diclofenac Sodium 3% gel - Test (Experimental): The diclofenac sodium 3% test gel is applied to lesion areas twice daily. It is to be smoothed onto the affected skin gently. The amount needed depends upon the size of the lesion site. Assure that enough Test Gel is applied to adequately cover each lesion. Normally 0.5 g of gel is used on each 5 cm x 5 cm lesion site.
  Interventions: Drug: Diclofenac sodium
- Diclofenac Sodium 3% gel - Reference (Active Comparator): The Reference diclofenac sodium 3% gel (Solaraze®) is applied to lesion areas twice daily. It is to be smoothed onto the affected skin gently. The amount needed depends upon the size of the lesion site. Assure that enough Reference (Solaraze®) Gel is applied to adequately cover each lesion. Normally 0.5 g of gel is used on each 5 cm x 5 cm lesion site.
  Interventions: Drug: Diclofenac sodium
- Placebo gel (Placebo Comparator): The placebo gel (contains no active ingredient) is applied to lesion areas twice daily. It is to be smoothed onto the affected skin gently. The amount needed depends upon the size of the lesion site. Assure that enough placebo gel is applied to adequately cover each lesion. Normally 0.5 g of gel is used on each 5 cm x 5 cm lesion site.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Diclofenac sodium — Topical administration of approximately 0.5g twice daily to the 25 sq cm treatment area for 60 days.
  Other Names: Solaraze
  Arms: Diclofenac Sodium 3% gel - Reference; Diclofenac Sodium 3% gel - Test
Other: Placebo — Topical administration of approximately 0.5g twice daily to the 25 sq cm treatment area for 60 days.
  Other Names: Vehicle base
  Arms: Placebo gel

SUMMARY:
To compare the relative efficacy and safety of the test formulation diclofenac sodium gel 3% (Actavis) to the marketed formulation Solaraze® (diclofenac sodium) Gel 3% (Fougera Pharms) in the treatment of the actinic keratosis

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form, which meets all criteria of current FDA and HIPAA regulations.
2. Immunocompetent male or non-pregnant, non-lactating female at least 18 years of age.
3. Diagnosis of AK with ≥ 5 and < 10 clinically typical, visible, discrete, nonhyperkeratotic, nonhypertrophic AK lesions each at least 4 mm in diameter on the face and/or bald scalp contained within a 25cm2 treatment area.
4. Women either must be 1 year post-menopausal (no menstrual periods for at least 12 months), surgically sterile, or if they are of child-bearing potential, they must:

   1. Have been using systemic birth control, IUD, or Norplant for at least 28 days prior to the start of treatment period of the study, or used barrier methods such as diaphragm plus spermicide or condom plus spermicide consistently, at least 14 days before study gel administration.
   2. Had a normal menstrual cycle for the month prior to the start of treatment.
   3. Have a negative urine pregnancy test result upon entry into the study.
   4. Agree to use a medically accepted form of birth control (oral, implant, injectable or transdermal contraceptives, intrauterine device, condom plus spermicide, diaphragm plus spermicide) or practice abstinence throughout the study period.
5. Free from any systemic or dermatologic disorder that, in the opinion of the Investigator, will interfere with the study results or increase the risk of AEs.
6. Any skin type or race, providing the skin pigmentation will allow discernment of erythema.
7. Willingness and capability to cooperate to the extent and degree required by the protocol.

Exclusion Criteria:

1. Active gastrointestinal ulceration or bleeding.
2. Current or history of severe renal or hepatic impairment.
3. Presence of atopic dermatitis, basal cell carcinoma, squamous cell carcinoma, eczema, psoriasis, rosacea, sunburn or other possible skin conditions on the face or bald scalp that in the investigator's opinion would interfere with the study assessments.
4. Use within six months prior to randomization of oral isotretinoin.
5. Use within six months prior to randomization on the face or bald scalp of 1) chemical peel, 2) dermabrasion, 3) laser abrasion, 4) PUVA (psoralen plus ultraviolet A) therapy, or 5) UVB therapy
6. Use within one month prior to randomization on the face or bald scalp of 1) cryodestruction or chemodestruction, 2)curettage, 3) photodynamic therapy, 4) surgical excision, 5)topical 5-fluorouracil, 6) topical corticosteroids, 7) topical diclofenac, 8) topical Imiquimod, 9) topical retinoids, or 10) other treatments for actinic keratosis including glycolic acids or over-the-counter products containing retinol, alpha or beta hydroxy acids.
7. Use within one month prior to randomization of 1)immunomodulators or immunosuppressive therapies, 2)interferon, 3) systemic corticosteroids or 4) cytotoxic drugs. (The occasional use of ophthalmic, nasal or inhaled steroids is acceptable and not reason for exclusion)
8. Known allergies to diclofenac sodium, benzyl alcohol, polyethylene glycol monomethyl ether 359, hyaluronate sodium or any excipients in the test or reference gels.
9. Receiving 5-Fluorouracil or other systemic cancer chemotherapy within 6 months prior to randomization.
10. Any condition, medical, psychological, or social, that, in the Investigator's opinion, would interfere with participation in the study.
11. Women who are pregnant, planning pregnancy or lactating.
12. Participation in any investigational drug study within 30 days of randomization or previous participation in this study.
13. Employees of the research center or Investigator.
14. Family members of employees of the research center or Investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 476 (Actual)
Dates: Start 2013-03; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry Lau, PhD, Study Director — Actavis Inc.
Locations (31):
- United States (31):
  - Investigator Site 23, Fremont, California
  - Investigator Site 9, Long Beach, California
  - Investigator Site 12, Newport Beach, California
  - Investigator Site 2, San Diego, California
  - Investigator Site 24, San Ramon, California
  - Investigator Site 14, Denver, Colorado
  - Investigator Site 17, Denver, Colorado
  - Investigator Site 21, Brandon, Florida
  - Investigator Site 25, Dunedin, Florida
  - Investigator Site 20, Fort Myers, Florida
  - Investigator Site 15, Jacksonville, Florida
  - Investigator Site 16, Miami, Florida
  - Investigator Site 6, Ormond Beach, Florida
  - Investigator Site 19, Winter Park, Florida
  - Investigator Site 22, Atlanta, Georgia
  - Investigator Site 11, Boise, Idaho
  - Investigator Site 8, Arlington Heights, Illinois
  - Investigator Site 28, Plainfield, Indiana
  - Investigator Site 31, Louisville, Kentucky
  - Investigator Site 27, Fridley, Minnesota
  - Investigator Site 13, Bozeman, Montana
  - Investigator Site 26, New Bern, North Carolina
  - Investigator Site 3, Raleigh, North Carolina
  - Investigator Site 18, Wilmington, North Carolina
  - Investigator Site 30, Cincinnati, Ohio
  - Investigator Site 1, Hazleton, Pennsylvania
  - Investigator Site 5, Clinton, South Carolina
  - Investigator Site 4, Johnson City, Tennessee
  - Investigator Site 10, Nashville, Tennessee
  - Investigator Site 7, West Jordan, Utah
  - Investigator Site 29, Midlothian, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Diclofenac Sodium 3% Gel: The test product diclofenac sodium 3% test gel is applied to lesion areas twice daily. It is to be smoothed onto the affected skin gently. The amount needed depends upon the size of the lesion site. Assure that enough Test Gel is applied to adequately cover each lesion. Normally 0.5 g of gel is used on each 5 cm x 5 cm lesion site.
  Diclofenac sodium: Topical administration of approximately 0.5g twice daily to the 25 sq cm treatment area for 60 days.
- Solaraze( Diclofenac Sodium) 3% Gel: The Reference diclofenac sodium 3% gel (Solaraze®) is applied to lesion areas twice daily. It is to be smoothed onto the affected skin gently. The amount needed depends upon the size of the lesion site. Assure that enough Reference (Solaraze®) Gel is applied to adequately cover each lesion. Normally 0.5 g of gel is used on each 5 cm x 5 cm lesion site.
  Diclofenac sodium: Topical administration of approximately 0.5g twice daily to the 25 sq cm treatment area for 60 days.
- Vehicle Gel: The vehicle (placebo) gel (contains no active ingredient) is applied to lesion areas twice daily. It is to be smoothed onto the affected skin gently. The amount needed depends upon the size of the lesion site. Assure that enough placebo gel is applied to adequately cover each lesion. Normally 0.5 g of gel is used on each 5 cm x 5 cm lesion site.
  Placebo: Topical administration of approximately 0.5g twice daily to the 25 sq cm treatment area for 60 days.
Period: Overall Study
Arm/Group | Diclofenac Sodium 3% Gel | Solaraze( Diclofenac Sodium) 3% Gel | Vehicle Gel
Started | 190 | 191 | 95
Completed | 160 | 163 | 83
Not Completed | 30 | 28 | 12
Not completed — Adverse Event | 4 | 4 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Non compliance with dosing requirements | 4 | 2 | 0
Not completed — Miscellaneous | 1 | 9 | 2
Not completed — Restricted medication | 5 | 1 | 1
Not completed — Serious Adverse Event | 1 | 0 | 0
Not completed — Withdrawal by Subject | 11 | 10 | 6
Not completed — Randomized in Error | 4 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Diclofenac Sodium 3% Gel | Solaraze( Diclofenac Sodium) 3% Gel | Vehicle Gel | Total
Number analyzed (Participants) | 188 | 189 | 93 | 470
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.34 (11.42) | 66.24 (11.37) | 65.55 (11.00) | 65.71 (11.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 54 | 26 | 136
  Male | 132 | 135 | 67 | 334
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 19 | 8 | 48
  Not Hispanic or Latino | 167 | 170 | 85 | 422
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 188 | 189 | 93 | 470
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With 100% Clearance of All AK Lesions Within the Treatment Area Assessed at Day 90
Description: The primary measure of bioequivalence will be evaluated using those patients who complete the study according to the (PP) population.
Time Frame: 90 days
Population: Analysis provided using the Per-Protocol Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Diclofenac Sodium 3% Gel | Solaraze( Diclofenac Sodium) 3% Gel | Vehicle Gel
Number analyzed (Participants) | 139 | 148 | 81
Participants
  Cure - 100% clearance of all AK lesions at Day 90 | 31 | 32 | 7
  No Cure - Not 100% Clearance of lesions at Day 90 | 108 | 116 | 74
Statistical Analysis 1: Comparison: Diclofenac Sodium 3% Gel vs Solaraze( Diclofenac Sodium) 3% Gel; Test type: Equivalence — 90% confidence interval of the difference in the percentage of patients between Test and Reference to be contained within -20%, + 20%, using the Per-Protocol Population; (Test-Ref) Difference = 0.68, 90% CI 2-sided [-8.06 to 9.42] — Applicable to Percentage of Subjects with Cure (100% complete AK clearance at day 90)
Statistical Analysis 2: Comparison: Diclofenac Sodium 3% Gel vs Vehicle Gel; Test type: Superiority; p = 0.0010, ANOVA

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Diclofenac Sodium 3% Gel | Solaraze( Diclofenac Sodium) 3% Gel | Vehicle Gel
All-Cause Mortality (participants affected / at risk) | 0/188 | 0/189 | 0/93
Serious Adverse Events (participants affected / at risk) | 7/188 | 4/189 | 2/93
Other Adverse Events (participants affected / at risk) | 102/188 | 91/189 | 35/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Diclofenac Sodium 3% Gel (N=188) | Solaraze( Diclofenac Sodium) 3% Gel (N=189) | Vehicle Gel (N=93)
Cardiac disorder (Cardiac disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0
Cardiac myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Alcoholism (Psychiatric disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Angioplasty (Surgical and medical procedures) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diclofenac Sodium 3% Gel (N=188) | Solaraze( Diclofenac Sodium) 3% Gel (N=189) | Vehicle Gel (N=93)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Bundle branch block right (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Mitral valce incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Cardiac disorders) | 1 (2) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye Swelling (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Periorbital oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoidal heamorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (3)
Oral discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Application site alopecia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Application site burn (General disorders) | 1 (1) | 0 (0) | 0 (0)
Application site dermatitis (General disorders) | 6 (6) | 3 (3) | 0 (0)
Application site dryness (General disorders) | 1 (1) | 0 (0) | 1 (2)
Application site exfoliation (General disorders) | 0 (0) | 3 (5) | 0 (0)
Application site haemorrhage (General disorders) | 0 (0) | 1 (1) | 0 (0)
Application site irritation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Application site pain (General disorders) | 2 (2) | 1 (1) | 2 (2)
Application site pruritus (General disorders) | 2 (2) | 2 (2) | 1 (1)
Application site rash (General disorders) | 1 (3) | 0 (0) | 0 (0)
Application site reaction (General disorders) | 1 (1) | 1 (1) | 0 (0)
Application site scab (General disorders) | 1 (3) | 0 (0) | 0 (0)
Application site swelling (General disorders) | 0 (0) | 3 (3) | 0 (0)
Application site urticaria (General disorders) | 0 (0) | 1 (1) | 0 (0)
Application site vesicles (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 2 (2) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 2 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Thirst (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 2 (2) | 0 (0) | 0 (0)
Acarodermatitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Application site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 3 (3)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastoenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Localized infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (3)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Respiratory rate decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cardiac myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Melanoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dementia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 5 (10) | 7 (9) | 3 (4)
Hyperaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Alcoholism (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 2 (4) | 0 (0)
Renal cyst (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary hypertention (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Sunburn (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Anal fissure excision (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Angioplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Malignant tumour excision (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Skin neoplasm excision (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Hypertention (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the study may be published or presented by the Investigator(s) after the review by, and in consultation and agreement with the Sponsor, and such that confidential or proprietary information is not disclosed.